CLINICAL TRIAL: NCT05172271
Title: A Feasibility Study of Transcranial Electric Stimulation Therapy (TEST) for Treatment Resistant Depression (TRD)
Brief Title: Transcranial Electric Stimulation Therapy (TEST) for Treatment Resistant Depression (TRD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: 210031; 21-M-0031
Record Dates: First submitted 2021-12-28; First posted 2021-12-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09-05

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Unipolar Major Depression
Keywords: Electroconvulsive Therapy; Major Depressive Disorder; noninvasive brain stimulation; Bipolar Disorder; SEIZURE
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Sham TEST (Sham Comparator): Anesthesia alone
  Interventions: Other: ECT device without stimulation
- Transcranial Electric Stimulation Therapy (TEST) (Experimental): TEST involves bifrontal electrical brain stimulation at a dose below the seizure threshold, applied in the same manner as standard electroconvulsive therapy (ECT), with scalp electrodes, under anesthesia, using a standard ECT device (modified or unmodified) that can deliver a range of doses below seizure threshold.
  Interventions: Device: MagPro TMS Stimulator and coil; Device: Thymatron(R) System IV; Device: Magnetic Resonance Imaging Scanner

INTERVENTIONS:
Device: MagPro TMS Stimulator and coil — TMS measurements of cortical excitability pre and post study intervention
  Arms: Transcranial Electric Stimulation Therapy (TEST)
Device: Thymatron(R) System IV — The Thymatron(R) System IV (Somatics LLC, Venice, FL, USA) is an FDA 510(k)-cleared ECT device. For TESt, we will be using it in a non FDA-approved manner--stimulating without intending to induce seizures.
  Arms: Transcranial Electric Stimulation Therapy (TEST)
Device: Magnetic Resonance Imaging Scanner — Conventional MRI studies in this protocol are considered non-significant risk (NSR) devices. While operated in research mode, the MRI will be under the International Electrotechnical Commission (IEC) 60601-2-33 First Level Controlled Operating Mode, which allows for research pulse sequences to be used within the FDA/IEC safety limits for MRI devices.
  Arms: Transcranial Electric Stimulation Therapy (TEST)
Other: ECT device without stimulation — Anesthesia alone
  Arms: Sham TEST

SUMMARY:
Background:

People with TRD are often helped by electroconvulsive therapy (ECT). But ECT can affect memory and thinking. Researchers want to study a treatment called TEST that uses less electricity.

Objective:

To study the safety and feasibility of TEST and assess its antidepressant effects.

Eligibility:

Adults aged 25-64 with major depression that has not been relieved by current treatments.

Design:

Participants will be admitted to the NIH Clinical Center for 5 18 weeks over 2 3 treatment phases. Their medications may be adjusted.

Participants will be interviewed about their depression, side effects, and other treatments they are receiving. They will complete questionnaires. They will give blood and urine samples. Their brain waves and heart rhythm will be recorded. They will take tests of memory, attention, mental functioning, and thinking.

Participants will have magnetic resonance imaging (MRI) scans of the head and brain. They will lie on a table that slides in and out of the scanner. Pictures of brain chemicals will also be taken. They may complete tasks during the MRI.

Participants will receive TEST and/or sham treatments. They may receive optional ECT. An intravenous catheter will be placed in an arm vein to receive general anesthesia. Two electrodes will be placed on the front of their head. An electric current will be passed from the ECT machine through the electrodes. For sham treatments, they will not receive the electric current. Their breathing, heart rate, brain function, blood pressure, and body movements will be measured.

Participants will have 7 follow-up visits over 6 months. Visits can be done via telehealth.

Participation will last for up to 42 weeks.

DETAILED DESCRIPTION:
Study Description:

This is a medical device feasibility study, which per FDA definition, is a study focusing primarily on continuing safety data collection that aims to capture preliminary safety and effectiveness data on a near-final or final device design to adequately plan an appropriate pivotal study. It tests the hypothesis that Transcranial Electric Stimulation Therapy (TEST), an experimental brain stimulation therapy, can have an antidepressant effect in individuals with treatment resistant depression (TRD) safely and without significant adverse cognitive effects. TEST involves bifrontal electrical brain stimulation at a dose below the seizure threshold, applied in the same manner as standard electroconvulsive therapy (ECT), with scalp electrodes, under anesthesia, using a standard ECT device. The effects of TEST will be compared to those of sham TEST (anesthesia alone) in 30 patients with TRD in a randomized, double-blind, parallel trial, followed by a nonrandomized extension during which all participants are eligible for active treatment.

Objectives:

Primary Objective: To evaluate the safety and feasibility of TEST in 30 adults with treatment resistant major depression (TRD)

Secondary Objectives: To assess the antidepressant effect of TEST.

Endpoints: Primary Endpoints: 1.Treatment adverse effects with an emphasis on adverse cognitive effects, primarily memory impairment. 2.Presence or absence of a seizure in participants receiving TEST (feasibility of consistently not inducing seizures with TEST)

Secondary Endpoint: Treatment-related changes in depressive symptom scale score

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of a signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, ages 25 through 64 years.
4. Meeting structured clinical interview for the DSM 5 (SCID) criteria for major depressive disorder, bipolar I disorder, or bipolar II disorder.
5. Currently have TRD as defined by a major depressive episode with lack of remission of depressive symptoms following two trials of different medication or one medication trial and one rTMS trial approved for unipolar or bipolar depression at adequate dosage and duration treatment consistent with an Antidepressant Treatment History Form (ATHF) confidence level >=3.
6. Score >= 25 on the Montgomery-Asberg Depression Rating Scale (MADRS) and a score >=2 on item 1 at screening or for individuals with bipolar depression, score >= 25 on the Bipolar Depression Rating Scale (BDRS) at screening.
7. Score <=12 on the Young Mania Rating Scale (YMRS) and a score <= 1 on item 1 at screening.
8. Willingness to: (a) provide written permission, as requested, to allow any and all forms of communication between the Investigator/Research Staff and any healthcare provider who currently provides and/or has provided service to the patient/subject within two years of study enrollment; and (b) provide the name and verifiable contact information of a person whom they trust to be an emergency contact whom research staff is at liberty to contact for the duration of study participation and who could serve as a legally authorized representative (LAR) if needed.
9. Agreement to remain on the same daily dose of all psychiatric medication(s) without taking any new psychiatric medication(s) for a minimum of 6 weeks (42 days) prior to the baseline assessment and through the completion of Study Phase III (Study Phase IV is the 6-month Follow-up Phase) unless advised otherwise by the Investigator
10. Agreement that dosage reduction of any medication taken for a psychiatric condition must be completed at least 4 weeks (28 days) prior to the baseline assessment and must remain unchanged thereafter through the completion of Study Phase III (Study Phase IV is the 6- month Follow-up Phase), unless advised otherwise by the Investigator
11. Agreement to remain on the same daily dose of psychiatric medication from the start of the baseline assessment / Phase I through the completion of the final treatment Study Phase III (Study Phase IV is the 6-month Follow-up Phase), unless advised otherwise by the Investigator.
12. For females of reproductive potential: use of contraception, which in the opinion of the Investigator is highly effective, for at least 1 month prior to screening and agreement to use such a method during study participation, except during the 6-month follow up.
13. Ability of the participant to understand and be willing to sign a written informed consent document as determined by the Investigator.

ECLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy or nursing or women planning to become pregnant during study period, except for the 6-month follow up phase.
2. A history of addiction to, dependence on, abuse of, or misuse of alcohol or any controlled, illicit, or illegal substance (excluding nicotine) within the past one year
3. Expression of recent or current active suicidal ideas and an explicit plan or intent, in the opinion of the Investigator or answering YES to questions 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) or scoring >4 on Montgomery-Asberg Depression Rating Scale (MADRS) item 10.
4. Presence of any disease, medical condition or physical condition that, in the opinion of the Investigator, may compromise, interfere with, limit, effect or reduce the:

   1. subject s ability to participate in any of the items listed in the Schedule of Activities
   2. integrity of the data or
   3. subject s ability to complete the full duration of the study.
5. Mood disorder is, in the opinion of the Investigator, significantly influenced or caused by an underlying medical or neurological condition, for example, multiple sclerosis or fibromyalgia
6. History of serious, potentially life-threatening reaction to methohexital or succinylcholine.
7. Clinically significant psychiatric comorbidity as determined by clinical interview and in the opinion of the Investigator
8. Past or present medical or neurological condition, disease, disorder or injury that, in the opinion of the Investigator, may significantly increase the potential risks of study participation, reduce or compromise a subject s ability to fully comply with all study requirements for the duration of the study or may compromise the integrity of the data. Past or present medical or neurological condition, disease, disorder or injury that, in the opinion of the Investigator, may significantly increase the potential risks of study participation, reduce or compromise a subject s ability to fully comply with all study requirements for the duration of the study or may compromise the integrity of the data.
9. History of seizure except those therapeutically induced by ECT, except for childhood febrile seizures.
10. History of any of the following:

    1. intracranial surgery
    2. cranial metal implants
    3. presence of devices that may be affected by MRI (pacemaker, medication pump, cochlear implant, implanted brain stimulator, vagus nerve stimulator
    4. history of head trauma associated with a brain imaging study that shows probable or definite evidence of a post-traumatic abnormality as determined by a neuroradiologist and which the Investigator deems clinically significant at screening.
11. Any of the following treatment histories:

    Failure to respond to adequate ECT treatment consistent with an ATHF confidence level >=3 in current or any previous episode

    Lifetime history of treatment with deep brain stimulation

    Use of any investigational drug or device within 4 weeks of the screening
12. Inability to pass the Evaluation to Sign A Consent Form test for adequate comprehension of the study for any reason including limitations related to use of the English language.
13. Positive HIV test.
14. Being an NIMH employee or an immediate family member of an NIMH employee.
15. Presence of any condition that, in the judgment of the investigator, may hinder completion of the procedures required by the study protocol.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Hopkins Verbal Learning Test-Revised (HVLT-R) | Baseline, End of Phase II (approximately 2 weeks) and end of Phase III (4-13 weeks) and at 2 and 4 weeks post treatment course
  The HVLT-R is a brief (<10 min) well-validated version of the word list delayed recall task that assesses anterograde memory.
change in EEG waveforms from pretreatment session baseline to end of treatment session | every treatment throughout course (approximately 3x weekly)
  This measure will determine the presence or absence of a seizure in participants receiving TEST. It will inform the feasibility of consistently not inducing seizures with TEST.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS), | Baseline, after every treatment (approximately 3x weekly) end of Phase II (approximately 2 weeks), end of Phase III (approximately 4-13 weeks), and during outpatient follow up every two weeks for the first month, then monthly for 5 months
  a 10-item, well validated, scale measuring depressive symptoms often used in ECT clinical trials.
Symptoms of Major Depressive Disorder Scale (SMDDS). | Baseline, after every treatment (approximately 3x weekly), end of Phase II (approximately 2 weeks), end of Phase III (approximately 4-13 weeks), and during outpatient follow up every two weeks for the first month, then monthly for 5 months
  The SMDDS is a 16-item, well validated, participant-administered scale that was developed to meet the recommendations promulgated by the FDA to guide industry in the conduct of depression clinical trials

CONTACTS AND LOCATIONS:
Overall Officials: William T Regenold, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants can opt in or out of our sharing their data and specimens w/othr researchers through the consent form. If participants opt in, our overall plan is to share a blood specimen and demographic (excluding PII) and clinical information that is deidentified and not linked to a code to which the sample or data can be traced for identification, with Gen ECT consortium which is part of the PGC. The samples and clinical information would be batched and sent once study data is reviewed and locked. Information to accompany the blood sample includes the following: 1. info about the blood sample-date collected 2. demographic information excluding PII 3. Clinical information and study results including the following: psychiatric and medical diagnoses; psychiatric and medical treatment history; substance use history; family history; reason for ECT, details of the ECT course, e.g., number of treatments, electrode placement, and results of cognitive testing and psychiatric scales.
Supporting Information: CSR
Time Frame: This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. @@@Data from this study may be requested from other (non-PGC) researchers indefinitely after the completion of the primary endpoint by contacting William T. Regenold, MDCM, Lead Associate Investigator. @@@Following publication of our study results, we will consider sharing deidentified clinical information and study results of individual participants as well as the study data analysis plan with potential collaborators who provide a methodologically sound proposal, as long as participants gave their permission at consent.
Access Criteria: IPD will be shared with potential collaborators who provide a methodologically sound proposal, and are willing to sign a data access agreement. The IPD can be used in any analyses, including meta-analyses, that are part of a methodologically sound proposal. The access mechanism will be through contacting study personnel listed in the clinicaltrials.gov study description or by directly contacting William T. Regenold, MDCM, Lead Associate Investigator. Requests will be reviewed by Dr. Regenold and the study PI, Dr. Sarah H. Lisanby.

REFERENCES:
- [Background] Prudic J, Sackeim HA, Devanand DP, Krueger RB, Settembrino JM. Acute cognitive effects of subconvulsive electrical stimulation. Convuls Ther. 1994 Mar;10(1):4-24. PMID 8055291
- [Background] Sackeim HA. Is the Seizure an Unnecessary Component of Electroconvulsive Therapy? A Startling Possibility. Brain Stimul. 2015 Sep-Oct;8(5):851-4. doi: 10.1016/j.brs.2015.07.026. Epub 2015 Jul 17. No abstract available. PMID 26358486
- [Background] Regenold WT, Noorani RJ, Piez D, Patel P. Nonconvulsive Electrotherapy for Treatment Resistant Unipolar and Bipolar Major Depressive Disorder: A Proof-of-concept Trial. Brain Stimul. 2015 Sep-Oct;8(5):855-61. doi: 10.1016/j.brs.2015.06.011. Epub 2015 Jun 26. PMID 26187603
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-M-0031.html